CLINICAL TRIAL: NCT03523572
Title: A Phase 1b, Multicenter, Two-Part, Open-Label Study of Trastuzumab Deruxtecan, an Anti-Human Epidermal Growth Factor Receptor-2 (HER2)-Antibody Drug Conjugate (ADC), in Combination With Nivolumab, an Anti-PD-1 Antibody, for Subjects With HER2-expressing Advanced Breast and Urothelial Cancer
Brief Title: Trastuzumab Deruxtecan With Nivolumab in Advanced Breast and Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Bristol-Myers Squibb (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U105; 2018-000371-32 (EudraCT Number)
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Urothelial Carcinoma
Keywords: Human epidermal growth factor receptor-2; HER2; Refractory; Metastatic; Urothelial cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Transitional Cell; Neoplasm Metastasis | interventions — trastuzumab deruxtecan; Nivolumab

STUDY DESIGN:
Intervention Model Description: Part 1 will be a sequential dose-finding (dose escalation) study, Part 2 will consist of a single group of four cohorts who receive the recommended dose (determined during Part 1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation (3.2 mg/kg) (Experimental): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 3.2 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
  The DLT observation period will be the first 2 cycles.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab
- Dose Escalation (5.4 mg/kg) (Experimental): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 3.2 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
  The DLT observation period will be the first 2 cycles.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab
- Dose Expansion - Cohort 1 (Experimental): Cohort 1: Participants with pathologically documented advanced/metastatic breast cancer that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines]. These participants received prior ado-trastuzumab emtansine (T-DM1).
  Participants will receive the RDE of trastuzumab deruxtecan and the flat dose of nivolumab.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab
- Dose Expansion - Cohort 2 (Experimental): Cohort 2: Participants with pathologically documented advanced/metastatic breast cancer that has centrally-determined low HER2 expression (IHC 1+ or IHC 2+/ISH-), who have exhausted treatments that can confer any clinically meaningful benefit (eg, other therapies such as hormonal therapy for patients who are hormone receptor positive).
  Participants received the RDE of trastuzumab deruxtecan and the flat dose of nivolumab.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab
- Dose Expansion - Cohort 3 (Experimental): Cohort 3: Participants with pathologically documented advanced/metastatic urothelial carcinoma that has centrally-determined HER2 expression of IHC 2+ or 3+, who received prior platinum-based therapy with documented progression.
  Participants received the RDE of trastuzumab deruxtecan and the flat dose of nivolumab.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab
- Dose Expansion - Cohort 4 (Experimental): Cohort 4: Participants with pathologically documented advanced/metastatic urothelial carcinoma that has centrally-determined HER2 expression of IHC 1+, who received prior platinum-based therapy with documented progression.
  Participants received the RDE of trastuzumab deruxtecan and the flat dose of nivolumab.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Nivolumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — The investigational product is a sterile lyophilized powder, which is made into solution for intravenous administration.
  Other Names: Enhertu®; T-DXd
Drug: Nivolumab — Nivolumab is an aqueous solution formulated at 10 mg/mL to be administered at a flat dose of 360 mg IV over 30 minutes. Protocol-defined thyroid testing is required while taking nivolumab.
  Other Names: Opdivo®

SUMMARY:
This is a study of trastuzumab deruxtecan for the treatment of HER2-positive unresectable or metastatic breast cancer following two or more prior anti-HER2 based regimens.

Participants will receive this study drug along with a cancer drug, an immune checkpoint inhibitor, anti-PD1, called nivolumab.

The study will be done in two parts:

* Part 1 is to identify the recommended dose to use for treatment.
* Part 2 is to find out how well the combination works, and how safe and tolerable it is.

DETAILED DESCRIPTION:
The purpose of this phase 1b (Part 1, Part 2) study is to assess the combination of a test drug (trastuzumab deruxtecan) with nivolumab in participants with HER2-expressing breast and urothelial cancer who had disease progression during or after prior therapies, did not respond to standard therapies, or for whom no standard therapy is available.

The study will be performed in 2 parts.

* Part 1 is to test different doses of trastuzumab deruxtecan when given along with a fixed dose of nivolumab, and establish the maximum tolerated dose/recommended dose for expansion, when used in combination with nivolumab
* Part 2 is to assess the efficacy and safety of this dose combination.

ELIGIBILITY:
Inclusion Criteria:

1. Is the age of majority (adulthood) in their country
2. Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1
3. Has pathologically documented breast cancer or urothelial cancer that is unresectable or metastatic, and refractory to or intolerant of existing therapy(ies) known to provide clinical benefit, and as specified in each study cohort
4. Has an adequate archival tumor sample available for the central laboratory to determine eligibility to participate
5. Has at least 1 measurable lesion per RECIST version 1.1
6. Has cardiac, bone marrow, kidney, liver, blood and clotting test results required per protocol
7. Has had an adequate washout period before enrollment since previous surgery and other treatment
8. If reproduction is possible, agrees to use protocol-defined methods of contraception (or completely abstain from heterosexual intercourse) from screening to at least 7 months for females and males after the last dose of study drug
9. Agrees to avoid harvesting sperm or ova for any reason from screening to at least 7 months for females and males after the last dose of study drug
10. Has a life expectancy of at least 3 months

Exclusion Criteria:

1. Has received prior treatment with nivolumab or trastuzumab deruxtecan
2. Has medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association classes II-IV). Troponin levels above upper limit of normal (ULN) at screening (as defined by the manufacturer) and without any MI-related symptoms should have a cardiologic consultation before enrollment to rule out MI.
3. Has a corrected QT interval by Fredericia (QTcF) prolongation to > 470 ms (females) or > 450 ms (males) based on an average of the screening triplicate 12-lead electrocardiogram
4. Has history of non-infectious interstitial lung disease (ILD/pneumonitis) (that required steroids), has ILD/pneumonitis currently, or it cannot be ruled out by imaging at screening
5. Has a condition (other than active autoimmune disease) that requires systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of starting study treatment
6. Is pregnant or breastfeeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (29):
- United States (10):
  - UCLA - Medical Center, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - University of Miami Hospital & Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Levine Cancer Institute Carolinas Healthcare System, Charlotte, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Tennessee Oncology - Sara Cannon Research Institute, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
- Belgium (3):
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
  - GZA Hospital Campus Sint-Augustinus, Wilrijk
- France (3):
  - Institut de Cancerologie de L'Ouest, Angers
  - Centre Georges Francois Leclerc, Dijon
  - ICO Rene Gauducheau, Saint-Herblain
- Germany (3):
  - Charite Campus Benjamin Franklin, Berlin, Brandenburg
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - University Cancer Center, Dresden, Saxony
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria Senese U.O.C. Immunoterapia Oncologica, Siena
- Spain (5):
  - Hospital Gregorio Maranon Madrid Spain, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramon y Cajal Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - START Madrid CIOCC, Madrid
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London, England
  - Royal Marsden Hospital (Surrey), Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 86 participants were enrolled and treated at 21 study sites in US and Europe. Final study results are reported for all outcome measures.
Pre-assignment Details: The Dose Escalation was intended to identify the maximum tolerated dose (MTD) of T-DXd in combination with a fixed dose of nivolumab.
Groups:
- Dose Escalation (3.2 mg/kg): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 3.2 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
- Dose Escalation (5.4 mg/kg): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
- Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines] and have received prior ado-trastuzumab emtansine (T-DM1) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined low HER2 expression (IHC 1+ or IHC 2+/ISH-) who have exhausted treatments that can confer any clinically meaningful benefit (e.g. other therapies such as hormonal therapy for patients who are hormone receptor positive) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC: Participants with pathologically documented advanced/metastatic urothelial carcinoma (UC) that has centrally-determined HER2 expression of IHC 2+ or 3+, who received prior platinum-based therapy with documented progression who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC: Participants with pathologically documented advanced/metastatic urothelial carcinoma (UC) that has centrally-determined HER2 expression of IHC 1+, who received prior platinum-based therapy with documented progression who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
Period: Dose Escalation
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) | Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Started (Only the Dose Escalation Phase is being presented.) | 4 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) | Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Started (Only the Dose Expansion Phase is being presented.) | 0 | 0 | 29 | 16 | 30 | 4
Completed | 0 | 0 | 6 | 1 | 4 | 0
Not Completed | 0 | 0 | 23 | 15 | 26 | 4
Not completed — Progressive Disease | 0 | 0 | 9 | 11 | 15 | 2
Not completed — Clinical Progression | 0 | 0 | 2 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 10 | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Full Analysis Set.
Groups:
- Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines] and have received prior ado-trastuzumab emtansine (T-DM1) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) | Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC | Total
Number analyzed (Participants) | 4 | 3 | 29 | 16 | 30 | 4 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 24 | 16 | 8 | 2 | 53
  >=65 years | 2 | 2 | 5 | 0 | 22 | 2 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.73 (10.978) | 63.99 (16.995) | 56.37 (9.799) | 48.11 (8.781) | 69.29 (10.352) | 59.71 (13.308) | 59.48 (12.672)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 29 | 16 | 27 | 3 | 82
  Male | 0 | 0 | 0 | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 5 | 0 | 0 | 0 | 6
  White | 3 | 3 | 23 | 14 | 28 | 4 | 75
  More than one race | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 2 | 0 | 3 | 2 | 7
  United States | 4 | 3 | 17 | 7 | 7 | 0 | 38
  Italy | 0 | 0 | 3 | 1 | 7 | 1 | 12
  United Kingdom | 0 | 0 | 3 | 1 | 1 | 0 | 5
  France | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Germany | 0 | 0 | 0 | 0 | 4 | 1 | 5
  Spain | 0 | 0 | 4 | 7 | 6 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities at 3.2 mg/kg and 5.4 mg/kg Dose Level in Participants With HER2-expressing Advanced Breast Cancer in Dose Escalation
Description: A Dose-Limiting Toxicity (DLT) is defined as any Treatment Emergent Adverse Event not attributable to disease or disease-related processes that occurs during the DLT evaluation period (2 complete cycles during Part 1) and is Grade 3 or above according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Each cycle is 21 days. Low dose was set at 3.2 mg/kg and high dose was set at 5.4 mg/kg.
Time Frame: Cycles 1 and 2 (each cycle is 21 days)
Population: DLT was assessed in the DLT evaluable set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Independent Central Review in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: The Objective Response Rate (ORR) was the defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by independent central review (ICR) committee based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on ICR is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: Every 6 weeks in the first year after Day 1 of Cycle 1 and thereafter every 12 weeks until disease progression or initiation of additional anticancer therapy and survival, up to 2 years 11.5 months (each cycle is 21 days)
Population: Objective response rate was assessed in the Full Analysis Set. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines] and have received prior ado-trastuzumab emtansine (T-DM1) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  The 3 participants enrolled in Dose Escalation (dosed at 5.4 mg/kg) were all HER2-positive and pooled with participants in Expansion Cohort 1 (5.4 mg/kg).
- Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC: Participants with pathologically documented advanced/metastatic urothelial carcinoma (UC) that has centrally-determined HER2 expression of IHC 1+, who received prior platinum-based therapy with documented progression who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  .
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 4 | 32 | 16 | 30 | 4
Percentage of Participants | 25.0 [NA to NA] — The curve that represents the upper CI for the response rate lies above 0.75, therefore the upper CI for first quartile could not be estimated. Similarly, the curve that represents the lower CI for the response rate lies above 0.75 and the lower CI for the quartile could not be estimated. | 65.6 [46.8 to 81.4] | 50.0 [24.7 to 75.3] | 36.7 [19.9 to 56.1] | 50.0 [NA to NA] — The curve that represents the upper CI for the response rate lies above 0.75, therefore the upper CI for first quartile could not be estimated. Similarly, the curve that represents the lower CI for the response rate lies above 0.75 and the lower CI for the quartile could not be estimated.

3. Secondary Outcome: Duration of Response (DoR) in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: Duration of Response (DoR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. DoR in participants with confirmed CR/PR based on independent central review and investigator assessment is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: Every 6 weeks in the first year after Day 1 of Cycle 1 and thereafter every 12 weeks until disease progression or initiation of additional anticancer therapy and survival, up to 5 years (each cycle is 21 days)
Population: Duration of Response (DoR) was assessed in the Full Analysis Set of participants with available data with confirmed CR/PR. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 0 | 44 | 15 | 23 | 3
months
  Independent Central Review: number analyzed (Participants) | 0 | 21 | 8 | 11 | 2
  Independent Central Review |  | NA [7.9 to NA] — Median was not reached at the end of follow up and the upper 95% CI was not estimable | 5.5 [2.8 to 8.0] | 13.1 [4.1 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated
  Investigator Assessment: number analyzed (Participants) | 0 | 23 | 7 | 12 | 1
  Investigator Assessment |  | 20.2 [10.4 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | 5.8 [5.2 to 10.4] | 8.7 [2.8 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated

4. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: Disease Control Rate (DCR) was defined as the percentage of participants who achieved a best overall response of CR, PR, or stable disease (SD) during study treatment. CR was defined as a disappearance of all target lesions, PR as at least a 30% decrease in the sum of diameters of target lesions, and SD as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Confirmation of CR/PR was required. DCR based on independent central review and investigator assessment is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: as for outcome 3
Population: Disease control rate was assessed in the Full Analysis Set. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 4 | 32 | 16 | 30 | 4
Percentage of Participants
  Independent Central Review | 50 [NA to NA] — There were not enough events to estimate a standard error for the DCR and the 95% CI could not be calculated | 93.8 [79.2 to 99.2] | 75.0 [47.6 to 92.7] | 76.7 [57.7 to 90.1] | 75.0 [NA to NA] — There were not enough events to estimate a standard error for the DCR and the 95% CI could not be calculated
  Investigator Assessment | 50 [NA to NA] — There were not enough events to estimate a standard error for the DCR and the 95% CI could not be calculated | 93.8 [79.2 to 99.2] | 87.5 [61.7 to 98.4] | 73.3 [54.1 to 87.7] | 50 [NA to NA] — There were not enough events to estimate a standard error for the DCR and the 95% CI could not be calculated

5. Secondary Outcome: Progression-Free Survival (PFS) in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: Progression-free survival (PFS) was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. PFS based on independent central review and investigator assessment is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: as for outcome 3
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 0 | 32 | 16 | 30 | 4
months
  Independent Central Review |  | 11.6 [6.9 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | 7.0 [2.3 to 10.8] | 6.9 [2.7 to 14.4] | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated.
  Investigator Assessment |  | 18.0 [11.0 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | 7.8 [2.4 to 9.8] | 5.5 [2.7 to 8.5] | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated.

6. Secondary Outcome: Time to Response (TTR) Based on Independent Central Review in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: Time to response (TTR) is defined as the time from the date of first dose of study treatment to the date of the first documented objective response (CR or PR). CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmation of CR/PR was required. TTR based on independent central review and investigator assessment is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: as for outcome 3
Population: Time to response was assessed in the Full Analysis Set. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 1 | 32 | 16 | 30 | 4
months | 1.41 [1.41 to 1.41] | 1.61 [1.2 to 5.5] | 3.73 [2.6 to 9.8] | 1.87 [1.2 to 6.9] | 3.25 [1.2 to 5.3]

7. Secondary Outcome: Overall Survival (OS) in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: Overall survival (OS) was defined as the time from the date of first dose of study drug to the date of death due to any cause. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: Date of first dose of study drug to the date of death due to any cause, up to 5 years
Population: Overall survival (OS) was assessed in the Full Analysis Set. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Escalation (3.2 kg/mg): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 3.2 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
Arm/Group | Dose Escalation (3.2 kg/mg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 4 | 32 | 16 | 30 | 4
months | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated | NA [20.8 to NA] — Median was not reached at the end of follow up and the upper 95% CI was not estimable | 19.5 [2.7 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | 11.0 [7.2 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it could not be calculated. | NA [NA to NA] — Median was not reached at the end of follow up and 95% CIs could not be calculated

8. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Investigator Assessment in Participants With HER2-expressing Advanced Breast Cancer or Urothelial Cancer
Description: The Objective Response Rate (ORR) was the defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigator assessment (IA) based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on IA is reported. As prespecified in the protocol, participants enrolled in Part 1 were pooled according to their trastuzumab deruxtecan dose and HER2 expressing levels (HER2 positive or HER2 low) for efficacy analyses. Participants who were dosed at 5.4 mg/kg of trastuzumab deruxtecan and have HER2-positive expression Breast Cancer (IHC score 3+ or IHC score 2+/ISH+) in Part 1 were pooled with the same participants from Part 2 (in this case, participants enrolled in Cohort 1).
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines] and have received prior ado-trastuzumab emtansine (T-DM1) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Includes 3 participants from Dose Escalation (5.4 mg/kg).
Arm/Group | Dose Escalation (3.2 kg/mg) | Dose Escalation (5.4 mg/kg) + Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 4 | 32 | 16 | 30 | 4
Percentage of Participants | 25 [NA to NA] — There were not enough events to estimate a standard error for the ORR and the 95% CI could not be calculated | 71.9 [53.3 to 86.3] | 43.8 [19.8 to 70.1] | 40.0 [22.7 to 59.4] | 25.0 [NA to NA] — There were not enough events to estimate a standard error for the ORR and the 95% CI could not be calculated

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after initiating the study drug until 47 days after last dose of study drug.
Time Frame: Date of signing the informed consent form up to 100 days after last dose of study drug or start of a new anticancer drug (whichever occurs first), up to 5 years
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation (5.4 mg/kg): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
Arm/Group | Dose Escalation (3.2 mg/kg) | Dose Escalation (5.4 mg/kg) | Dose Expansion Cohort 1 (5.4 mg/kg): HER2 Positive BC | Dose Expansion Cohort 2 (5.4 mg/kg): HER2 Low BC | Dose Expansion Cohort 3 (5.4 mg/kg): HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4 (5.4 mg/kg): HER2 Low Expressing (IHC 1+) UC
Number analyzed (Participants) | 4 | 3 | 29 | 16 | 30 | 4
Participants | 4 | 3 | 29 | 16 | 30 | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 100 days after last dose of the study drug, up 5 years.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Groups:
- Dose Escalation (3.4 mg/kg): Participants with HER2-expressing breast cancer who received starting intravenous dose of trastuzumab deruxtecan at 3.2 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
  Escalating/de-escalating doses of trastuzumab deruxtecan in combination with a flat dose of nivolumab was administered on Day 1 of each 21-day cycle.
- Dose Expansion Cohort 1: HER2 Positive BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined positive HER2 expression (IHC 3+ or IHC 2+/ISH+) [as defined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines] and have received prior ado-trastuzumab emtansine (T-DM1) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 2: HER2 Low BC: Participants with pathologically documented advanced/metastatic breast cancer (BC) that has centrally-determined low HER2 expression (IHC 1+ or IHC 2+/ISH-) who have exhausted treatments that can confer any clinically meaningful benefit (e.g. other therapies such as hormonal therapy for patients who are hormone receptor positive) who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 3: HER2 High Expressing (IHC 2+/3+) UC: Participants with pathologically documented advanced/metastatic urothelial carcinoma (UC) that has centrally-determined HER2 expression of IHC 2+ or 3+, who received prior platinum-based therapy with documented progression who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
- Dose Expansion Cohort 4: HER2 Low Expressing (IHC 1+) UC: Participants with pathologically documented advanced/metastatic urothelial carcinoma (UC) that has centrally-determined HER2 expression of IHC 1+, who received prior platinum-based therapy with documented progression who received starting intravenous dose of trastuzumab deruxtecan at 5.4 mg/kg and a fixed intravenous dose of 360mg of nivolumab every 3 weeks (Q3W).
Arm/Group | Dose Escalation (3.4 mg/kg) | Dose Escalation (5.4 mg/kg) | Dose Expansion Cohort 1: HER2 Positive BC | Dose Expansion Cohort 2: HER2 Low BC | Dose Expansion Cohort 3: HER2 High Expressing (IHC 2+/3+) UC | Dose Expansion Cohort 4: HER2 Low Expressing (IHC 1+) UC
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/3 | 7/29 | 8/16 | 17/30 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 12/29 | 4/16 | 17/30 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 29/29 | 16/16 | 30/30 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation (3.4 mg/kg) (N=4) | Dose Escalation (5.4 mg/kg) (N=3) | Dose Expansion Cohort 1: HER2 Positive BC (N=29) | Dose Expansion Cohort 2: HER2 Low BC (N=16) | Dose Expansion Cohort 3: HER2 High Expressing (IHC 2+/3+) UC (N=30) | Dose Expansion Cohort 4: HER2 Low Expressing (IHC 1+) UC (N=4)
Disease Progression (General disorders) | 0 | 1 | 1 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Postprocedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Troponin T Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urostomy Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation (3.4 mg/kg) (N=4) | Dose Escalation (5.4 mg/kg) (N=3) | Dose Expansion Cohort 1: HER2 Positive BC (N=29) | Dose Expansion Cohort 2: HER2 Low BC (N=16) | Dose Expansion Cohort 3: HER2 High Expressing (IHC 2+/3+) UC (N=30) | Dose Expansion Cohort 4: HER2 Low Expressing (IHC 1+) UC (N=4)
Nausea (Gastrointestinal disorders) | 2 | 1 | 16 | 10 | 22 | 3
Fatigue (General disorders) | 1 | 3 | 14 | 6 | 16 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 9 | 8 | 14 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 11 | 6 | 13 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 14 | 7 | 8 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 11 | 6 | 12 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 11 | 8 | 8 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 13 | 6 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 6 | 6 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 5 | 0 | 11 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 7 | 4 | 4 | 0
Oedema Peripheral (General disorders) | 3 | 2 | 6 | 2 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 3 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 4 | 2 | 1
Headache (Nervous system disorders) | 1 | 0 | 4 | 3 | 5 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 4 | 2 | 5 | 1
Vision Blurred (Eye disorders) | 1 | 0 | 8 | 1 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 3 | 2 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 5 | 3 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 6 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 1 | 4 | 2
Pyrexia (General disorders) | 1 | 0 | 5 | 1 | 5 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 2 | 3 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 6 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 2 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 4 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 4 | 2 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 6 | 2
Neutrophil Count Decreased (Investigations) | 0 | 0 | 3 | 2 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 4 | 3 | 1 | 1
Amylase Increased (Investigations) | 1 | 0 | 4 | 2 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 4 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 6 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 4 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 3 | 0
Dry Eye (Eye disorders) | 1 | 0 | 3 | 2 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 2 | 3 | 1
Lipase Increased (Investigations) | 1 | 0 | 2 | 0 | 4 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 3 | 2 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 1 | 2 | 2 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 3 | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 2 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0 | 3 | 0 | 2 | 0
Disease Progression (General disorders) | 0 | 1 | 1 | 1 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 4 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 0
Malaise (General disorders) | 0 | 0 | 3 | 1 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 3 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 1 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Lethargy (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Otitis Media (Ear and labyrinth disorders) | 1 | 0 | 2 | 0 | 0 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Renal Pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Addison's Disease (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bilirubin Conjugated Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Bilirubin Unconjugated Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eyelid Skin Dryness (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Folate Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hernia Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retinal Tear (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Mood Altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03523572/Prot_SAP_000.pdf